CLINICAL TRIAL: NCT05582096
Title: A Dose-Escalation Treatment, Phase 1, Investigator- and Participant-Blind, Placebo-controlled Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of LY3457263 in Combination With Tirzepatide in Overweight or Obese Participants
Brief Title: A Study of LY3457263 in Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18463; J1R-MC-GZFC (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3457263 + Tirzepatide (Experimental): LY3457263 administered subcutaneously (SC) in combination with tirzepatide given SC.
  Interventions: Drug: LY3457263; Drug: Tirzepatide
- Placebo + Tirzepatide (Placebo Comparator): Placebo administered SC in combination with tirzepatide given SC.
  Interventions: Drug: Tirzepatide; Drug: Placebo

INTERVENTIONS:
Drug: LY3457263 — Administered SC.
  Arms: LY3457263 + Tirzepatide
Drug: Tirzepatide — Administered SC.
  Other Names: LY3298176
Drug: Placebo — Administered SC.
  Arms: Placebo + Tirzepatide

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3457263 when administered in combination with tirzepatitide in overweight or obese participants. The study will also evaluate how much of LY3457263 gets into the blood stream and how long it takes the body to remove it in overweight or obese participants. The study will last up to approximately 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Have a stable body weight and body mass index (BMI) within the range 27.0 to 45.0 kilograms per meter squared (kg/m²)
* Male or female participants not of childbearing potential

Exclusion Criteria:

* Have a mean sitting systolic blood pressure (BP) higher than 160 millimeters of mercury (mmHg) or a mean sitting diastolic BP higher than 90 mmHg from 3 measurements
* Have an abnormal 12-lead electrocardiogram (ECG) at screening
* Have type 1 or type 2 diabetes mellitus

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to 11 weeks
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3457263 | Predose on Day 1 up to 43 days postdose
  PK: AUC of LY3457263

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- LabCorp CRU, Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No